CLINICAL TRIAL: NCT05013437
Title: A Pilot Study to Assess Impact of Low Dose Melphalan on Disease Burden Measured by Next Generation Sequencing Before Autologous Hematopoietic Cell Transplant (AHCT) for Multiple Myeloma Patients
Brief Title: Melphalan on Disease Burden Measured by Next Generation Sequencing Before AHCT (Autologous Hematopoietic Cell Transplant) for Multiple Myeloma
Acronym: AHCT
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The original principal Investigator left the institution.
Sponsor: Koen van Besien (Other)
Responsible Party: Sponsor-Investigator, Koen van Besien, MD, PhD, Division Chief, Hematology and Cellular Therapy, UH Cleveland Medical Center, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1A20
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; High-Throughput Nucleotide Sequencing; Prochlorperazine; Acetaminophen; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Evomela (Melphalan) (Experimental): Participants will receive Evomela 16 mg/m2 on day 1 of the study only. Evomela will be given as IV infusion over 30 minutes after administration of 500 cc normal saline as pre-hydration and pre-medications Prochlorperazine, Acetaminophen, and Diphenhydramine.
  Interventions: Drug: Evomela; Device: Next Generation Sequencing; Drug: Prochlorperazine; Drug: Acetaminophen; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Evomela — 16 mg/m^2 Evomela administered one time via a central line
  Other Names: Melphalan
Device: Next Generation Sequencing — Next Generation Sequencing
Drug: Prochlorperazine — 10mg once intravenous (IV) within 30 minutes before Evomela
Drug: Acetaminophen — 650 mg once orally within 30 minutes before Evomela
Drug: Diphenhydramine — 50 mg once intravenously within 30 minutes before Evomela

SUMMARY:
The purpose of this study is to see if Multiple Myeloma (MM) cells are sensitive to the chemotherapy used in transplant or not. The main chemotherapy agent utilized in stem cell transplant is melphalan. The study will utilize 1/10 of the dose used in transplant to study sensitivity of the tumor to melphalan. Melphalan is approved by the U.S. Food and Drug Administration (FDA) for transplant for MM patients.

DETAILED DESCRIPTION:
Currently, there is no method to predict whether a patient will have benefit from stem cell transplant or not. The usual approach is to proceed to stem cell transplant as long as a patient with MM has adequate organ function, meaning heart, kidney, lungs and other organs can tolerate the complications from transplant.

In this study, all participants will already have had pre-collection bone marrow aspirate as standard of care that will be available for minimal residual disease (MRD) testing by NGS platform. Participants will receive only one, low-dose of melphalan (Evomela) intravenously. Participants will be asked to return to clinic for a follow-up visit at one week and two weeks after the infusion. Another bone marrow aspirate will be performed after 2 weeks from the day of Evomela administration. After the study, participants will have a standard-of-care (SOC) autologous stem cell transplant.

The primary objective is to evaluate the impact of a test dose of low dose melphalan (16 mg/m2) before autologous hematopoietic cell transplant on disease volume measured by Next Generation Sequencing (NGS).

Secondary objectives are:

* To assess safety of low dose melphalan after CD34 (cluster of differentiation 34) collection and before high-dose melphalan-based autologous stem cell transplant.
* To describe the impact of a test dose of low dose melphalan (16 mg/m2) before autologous hematopoietic cell transplant on disease volume measured by peripheral blood Mass Spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have diagnosis of symptomatic MM
* Participants must have received at least three cycles of anti-myeloma regimen including a proteasome inhibitor (i.e., bortezomib, carfilzomib or ixazomib) plus Lenalidomide or daratumumab, and have future plan of autologous stem cell transplant.
* Participants must have achieved Partial Response based on International Myeloma Working Group response criteria (Appendix II).
* Participants must have at least equal or greater than 100 mg/dL or 0.1 gr/dL monoclonal protein on serum electrophoresis and immunofixation at diagnosis
* Minimum 3 x10^6/kg collected CD34+cells in one or multiple days. (CD=cluster of differentiation)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2. Life expectancy ≥ 12 months
* Adequate hepatic function, as defined by:

  * Serum ALT ≤ 3.5 times the upper limit of normal (ALT=alanine aminotransferase)
  * Serum direct bilirubin ≤ 2 mg/dL (34 μmol/L) within 21 days prior to initiation of therapy
* Creatinine clearance (CrCl) ≥ 40 mL/minute within 21 days prior to start of therapy either measured or calculated using a standard formula (e.g., Cockcroft and Gault).
* Adequate bone marrow function ,as defined by:

  * Hemoglobin ≥ 10.0 g/dl
  * WBC (white blood cell count) ≥ 3.00 x 10^9/L
  * Absolute neutrophil count ≥1.5 x10^9/L
  * Platelets ≥ 100 x 10^9/L ---Growth factors are not allowed to be used in order to meet adequate bone marrow function
* Written informed consent in accordance with federal, local, and institutional guidelines
* Participants of childbearing potential must agree to practice reliable contraception for at least 28 days before and for 60 days after last dose of study drug. Reliable contraception is defined as:

  * One highly effective method and one additional effective (barrier) method:

    * Examples of highly effective methods:

      * Intrauterine device (IUD)▪Hormonal (injections, implants, levonorgestrel releasing intrauterine system [IUS], medroxyprogesterone acetate depot injections, ovulation inhibitory progesterone-only pills [e.g.desogestrel])
      * Tubal ligation
      * Partner's vasectomy
    * Examples of additional effective methods

      * Male condom
      * Diaphragm
      * Cervical Cap

Exclusion Criteria:

* Prior treatment toxicities have not resolved to ≤ Grade 2 according to NCI CTCAE Version 5.0 (except neuropathy).
* Participant receiving any other investigational agents within 21 days prior to study/treatment
* Treatment with any anti-myeloma chemotherapy within 14 days
* Diagnosis of amyloidosis, POEMS.
* Major surgery, radiotherapy or infection requiring therapy within 14 days of starting study treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to melphalan
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because melphalan is an alkalizing agent with the potential for teratogenic or abortifacient effects. Because there is unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with melphalan, breastfeeding should be discontinued if the mother is treated with melphalan
* Unstable angina or myocardial infarction within 4 months prior to registration, NYHA (New York Heart Association) Class II, III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker.
* Cerebrovascular disease manifested as prior stroke at any time or TIA (transient ischemic attack) in the 12 months prior to initiation of therapy
* Non-hematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b)carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas.
* Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Residual myeloma cell number measured by NGS | At baseline
  Myeloma disease response will be assessed by residual myeloma cell number measured via NGS method, utilizing clonoSEQ (assay) before and after low dose Evomela. The clonoSEQ Assay measures minimal residual disease (MRD) to monitor changes in burden of disease during and after treatment. MRD refers to the number of MM cells that remain in a person during and following treatment.
Residual myeloma cell number measured by NGS | After treatment, day 15
  Myeloma disease response will be assessed by residual myeloma cell number measured via NGS method, utilizing clonoSEQ before and after low dose Evomela. The clonoSEQ Assay measures minimal residual disease (MRD) to monitor changes in burden of disease during and after treatment. MRD refers to the number of MM cells that remain in a person during and following treatment.

SECONDARY OUTCOMES:
Toxicity in pre-transplant period assessed according to CTCAE v. 5.0 | Days 1, 8, 15, and 52
  Toxicity in pre-transplant period assessed according to Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0.
Percent of participants with pre-transplant period safety | Days 1, 8, 15, and 52
  Safety will be assessed by absence of any grade 4 or 5 clinically relevant therapy-related toxicity, or grade 3 clinically significant, therapy-related toxicities that do not resolve to grade ≤ 2 within one week
Percent of participants with diarrhea and oral mucositis and other non-hematologic toxicities | Day 52
  Percent of participants with diarrhea and oral mucositis and other non-hematologic toxicities will be assessed according to CTCAE v.5.0 during the inpatient transplant phase.
Percent of participants with post-transplant period safety | Day 52
  Safety assessed by absence of any grade 4 or higher diarrhea or oral mucositis lasting more than 2 days.
Percent of participants with engraftment failure | Day 52
  Neutrophil engraftment will be defined as the first day of 3 consecutive lab values obtained on different days when the ANC (absolute neutrophil count) is greater than or equal to 0.5 x 109/L (500/μl). Any Engraftment later than 28 days after hematopoietic stem cell infusion will count as engraftment failure.
Percent of participants with safety stopping endpoints | Day 52
  The following study drug-related toxicities, assessed based on CTCAE v.5.0, will count as safety stopping endpoints for this trial:
  1. non-hematologic toxicity grade 3 or higher that do not resolve to ≤grade 2 within one week occurring in any patient at any time during the study;
  2. any grade 4 toxicity in two or more patients with any duration in the pre-transplant phase and
  3. any oral mucositis or diarrhea grade 4 toxicity in two or more patients last more than 2 days in the inpatient transplant phase.
  4. Neutrophil engraftment failure in more than 2 patients (10% of enrolled patients), and
  5. any death on trial whether in pre-transplant or post-transplant phase.

CONTACTS AND LOCATIONS:
Overall Officials: Koen van Besien, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in publication
Supporting Information: Study Protocol, SAP, CSR